CLINICAL TRIAL: NCT06404801
Title: Development of Stance Control Orthotic Knee Joint For Improvement of KAFO Users
Status: Active, not recruiting | Type: Observational
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Other Study IDs: MSRSW/Batch-Fall22/706
Record Dates: First submitted 2024-05-05; First posted 2024-05-08 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Ankle Osteoarthritis; Knee

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Stance Control — Instead of stability coming from a locked knee joint, the brace is able to lock and unlock at just the right time while walking

SUMMARY:
I want to design Stance control orthotic knee joint for improvement of KAFO users which is not available in Pakistan imported stance control orthotic knee joints are very expensive patients can't afford. The aim of my study to develop low cost stance control knee joint and ensure its availablity for KAFO users.

ELIGIBILITY:
Inclusion Criteria:

* Polio Patient
* Proximal tibial fracture.

Exclusion Criteria:

* Patients without KAFO
* Cerebral Palsy Patients

Ages: 16 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: peoples selected based on having Polio or Proximal tibial fracture
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Patient Satisfaction Through Questionnaire | 12 Months
  Through Questionnaire used to ask after the use of stance control to messure the pain in the pionts used in questioner
SF-36 | 12 months
  physical functioning (PF), role physical (RP), bodily pain (BP), general health (GH), vitality (VT), social functioning (SF), role emotional (RE), and mental health (MH)

CONTACTS AND LOCATIONS:
Locations (1):
- Peshawar North West General Hospital & Research Center, Peshawar, Khyber Pakhtunkhwa, Pakistan

IPD SHARING:
Plan to Share IPD: No